CLINICAL TRIAL: NCT02282722
Title: Improving Informed Consent for Palliative Chemotherapy: Development of a Regimen-Specific Multi-Media Informed Consent Library To Promote Patient-Centered Decision-Making About Treatment of Advanced Gastrointestinal Cancers
Brief Title: Improving Informed Consent for Palliative Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Alliance for Clinical Trials in Oncology (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrea Enzinger, Chief, Division of Population Sciences, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-143; CE-1304-6517 (Other Grant/Funding Number: PCORI); 1UG1CA189823-01 (NIH)
Record Dates: First submitted 2014-10-27; First posted 2014-11-04 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Pancreatic Cancer; Unresectable Pancreatic Cancer
Keywords: cancer; palliative; chemotherapy; metastatic; colorectal; communication; informed consent; video; education; oncology; patient-centered; outcomes research
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Neoplasms; Neoplasm Metastasis; Communication | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual informed consent (Active Comparator): Study participant will receive usual, standard-of-care informed consent for chemotherapy materials.
  Interventions: Other: Usual, standard-of-care informed consent for chemotherapy
- Investigational informed consent (Experimental): Study participant will receive investigational informed consent for chemotherapy materials that were developed by the study team.
  Interventions: Other: Investigational informed consent for chemotherapy

INTERVENTIONS:
Other: Investigational informed consent for chemotherapy — Investigational informed consent materials consist of regimen-specific multimedia tools: a video plus a booklet.
  Arms: Investigational informed consent
Other: Usual, standard-of-care informed consent for chemotherapy — The enrolling site's institutional standard-of-care informed consent materials.
  Arms: Usual informed consent

SUMMARY:
Patients are routinely asked to sign an "informed consent" document prior to starting chemotherapy, indicating they understand the risks and benefits of treatment. Although this could be a strategic moment to equip patients with information they need to make truly informed medical decisions, many patients and caregivers note that these conversations are less useful than they could be. The informed consent process and its associated documents suffer several limitations: 1) risks are emphasized over benefits; 2) educational materials focus on individual drugs instead of regimens; 3) information is presented in written instead of alternative written/audiovisual format; and 4) the patient perspective is lacking.

The overarching objective of this project is to develop a library of communication tools for the most common chemotherapy regimens used to treat advanced gastrointestinal cancers. Tools will include video clips and written documents that can be readily distributed, modified, and customized. This toolkit will be crafted in collaboration with oncologists and patients living with gastrointestinal cancer and improves upon existing resources in several ways: 1) balanced discussion of benefits as well as risks, 2) focus on regimens rather than drugs, 3) use of both written and video format, and 4) inclusion of the patient perspective (e.g. video clips of patients describing their experience). A panel of oncologist and patient stakeholders will evaluate the acceptability of the tools. The investigators will then conduct a randomized clinical trial to demonstrate if the informed consent toolkit improves the quality of informed consent for palliative chemotherapy. If effective, the tools will be amenable to broad dissemination via patient accessible cancer education websites and oncology clinics.

DETAILED DESCRIPTION:
Research indicates that many patients with advanced cancer receive palliative chemotherapy without sufficient understanding of its likely risks and benefits. In surveys, many patients receive palliative chemotherapy without expressing an understanding that cure is unlikely.

The root of this problem is undoubtedly complex, but may relate to gaps in communication and patient education about the risks and benefits of treatment. Patients are routinely asked to sign an "informed consent" document prior to starting chemotherapy, indicating they understand the risks and benefits of treatment. Although this could be a strategic moment to equip patients with information they need to make truly informed medical decisions, many patients and caregivers note that these conversations are less useful than they could be. The informed consent process and its associated documents suffer several limitations: 1) risks are emphasized over benefits; 2) educational materials focus on individual drugs instead of regimens; 3) information is presented in written instead of alternative written/audiovisual format; and 4) the patient perspective is lacking.

The overarching objective of this trial is to test a suite of patient-centered videos and booklets to support informed consent for common chemotherapy regimens used to treat advanced gastrointestinal cancers. In this study, patients with metastatic colorectal cancer, locally advanced and metastatic pancreatic cancer considering treatment with first or second-line palliative chemotherapy were randomized to the usual process of chemotherapy informed consent, or usual care supplemented by access to the appropriate investigational chemotherapy informed consent video and booklet. Patients were surveyed at baseline, 2-weeks post-treatment initiation, and 3 months regarding their understanding of chemotherapy risks and benefits, decisional conflict, and other metrics of informed decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced colorectal cancer with metastasis, locally advanced pancreatic cancer, or metastatic pancreatic cancer.
* Is considering treatment with 1st line or 2nd line chemotherapy
* Treating oncologist has recommended consideration of one or more of the regimens for which we have developed informed consent materials
* Age ≥ 21
* English proficiency (reading and speaking)

Exclusion Criteria:

* Significant delirium/dementia as judged by the treating physician
* Isolated liver metastases being evaluated for curative resection

In addition, caregivers of eligible patients will also be eligible to participate in the caregivers assessments.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - University of California at San Francisco, San Francisco, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber at Milford, Milford, Massachusetts
  - Dana-Farber at South Shore, South Weymouth, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health, Winston-Salem, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
If interested in obtaining data from this project, please contact PI Deb Schrag at deb_schrag@dfci.harvard.edu.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available after the completion of primary outcome analyses and for up to 10 years following.
Access Criteria: If interested in obtaining data from this project, please contact PI Deb Schrag at deb_schrag@dfci.harvard.edu.

REFERENCES:
- [Background] Weeks JC, Catalano PJ, Cronin A, Finkelman MD, Mack JW, Keating NL, Schrag D. Patients' expectations about effects of chemotherapy for advanced cancer. N Engl J Med. 2012 Oct 25;367(17):1616-25. doi: 10.1056/NEJMoa1204410. PMID 23094723
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Background] Mazor KM, Street RL Jr, Sue VM, Williams AE, Rabin BA, Arora NK. Assessing patients' experiences with communication across the cancer care continuum. Patient Educ Couns. 2016 Aug;99(8):1343-8. doi: 10.1016/j.pec.2016.03.004. Epub 2016 Mar 6. PMID 26979476
- [Background] Legare F, Kearing S, Clay K, Gagnon S, D'Amours D, Rousseau M, O'Connor A. Are you SURE?: Assessing patient decisional conflict with a 4-item screening test. Can Fam Physician. 2010 Aug;56(8):e308-14. PMID 20705870
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Derived] Enzinger AC, Uno H, McCleary N, Frank E, Sanoff H, Van Loon K, Matin K, Bullock A, Cronin C, Cibotti H, Bagley J, Schrag D. Effectiveness of a Multimedia Educational Intervention to Improve Understanding of the Risks and Benefits of Palliative Chemotherapy in Patients With Advanced Cancer: A Randomized Clinical Trial. JAMA Oncol. 2020 Aug 1;6(8):1265-1270. doi: 10.1001/jamaoncol.2020.1921. PMID 32672806

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 216 participants were consented to this study. Of these, 16 were were not eligible to be randomized and 14 did not complete a baseline assessment. After consultations with the study statistician, these participants were intentionally excluded from our analytic cohort. Therefore, 186 participants are included in the participant flow module.
Groups:
- Patient Usual Care Arm: Patients randomized to usual care informed consent materials.
- Patient Investigational Care Arm: Patients randomized to the investigational informed consent materials.
Period: Overall Study
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
Started | 94 | 92
2-week Assessment | 79 | 75
3-month Assessment | 71 | 73
Completed | 71 | 73
Not Completed | 23 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Informed Consent | Investigational Informed Consent | Total
Number analyzed (Participants) | 94 | 92 | 186
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 56 | 113
  >=65 years | 37 | 36 | 73
Age, Continuous [Mean (Full Range); unit: Years] | 59.2 [30 to 85] | 59.4 [28 to 86] | 59.3 [28 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 39 | 79
  Male | 54 | 53 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 6 | 17
  White | 76 | 84 | 160
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Live alone [Count of Participants; unit: Participants]
  Yes | 16 | 12 | 28
  No | 76 | 79 | 155
  Unknown | 2 | 1 | 3
Education [Count of Participants; unit: Participants]
  Grade school or less | 8 | 5 | 13
  High school graduate, or some college | 36 | 29 | 65
  College degree or higher | 49 | 57 | 106
  Unknown/missing | 1 | 1 | 2
Diagnosis [Count of Participants; unit: Participants]
  Metastatic colorectal cancer | 59 | 59 | 118
  Advanced pancreatic cancer | 35 | 33 | 68
ECOG Performance Status [Count of Participants; unit: Participants]
  0 - Fully Active | 31 | 44 | 75
  1 - Restricted in physically strenuous activity | 42 | 26 | 68
  2 - Ambulatory but unable to work | 5 | 6 | 11
  3 - Capable of limited self-care | 0 | 0 | 0
  4 - Completely disabled | 0 | 0 | 0
  Unknown/Missing | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Accurate Understanding of Chemotherapy Benefits
Description: Patients were asked "How likely do you think that chemotherapy is to cure your cancer?" with response options of not at all likely, a little likely, somewhat likely, very likely, and don't know. A response of "not at all likely" was considered accurate. All other responses, including don't know, were considered inaccurate.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
Number analyzed (Participants) | 71 | 73
Participants
  Accurate | 39 | 39
  Inaccurate | 30 | 31
  Did not answer | 2 | 3

2. Secondary Outcome: Number of Patients With Accurate Understanding of Chemotherapy Risks
Description: Patients were asked to rate the likelihood that they would experience specific side effects as a result of the chemotherapy under consideration, with separate items for nausea/vomiting, diarrhea, neuropathy, and hair loss. Patients' responses were correlated to the known side effect profile of their chemotherapy regimen and coded as accurate or inaccurate.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
Number analyzed (Participants) | 79 | 75
Participants
  Inaccurate | 47 | 33
  Accurate | 31 | 41
  Unknown/missing | 1 | 1

3. Secondary Outcome: Number of Participants With Accurate Understanding of the Goals of Palliative Chemotherapy
Description: Patients were asked "according to your doctor, what is the goal of the chemotherapy?" with the ability to choose any/all of the following response options: cure, control cancer growth, alleviate symptoms, prolong life, or other. Selecting either control cancer growth, and/or alleviate symptoms, and/or prolong life were defined as accurate understanding; "to cure" was considered inaccurate.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
Number analyzed (Participants) | 79 | 75
Participants
  Inaccurate | 10 | 9
  Accurate | 68 | 65
  Unknown/missing | 1 | 1

4. Secondary Outcome: Decisional Conflict When Making a Chemotherapy Treatment Choice: Modified SURE Scores
Description: Decisional Conflict was assessed by a modified version of the 4 item SURE instrument of Legare at al which assesses whether patients 1) are sure of the best treatment option, 2) know the risks and benefits of their treatment options, 3) are clear about which risks and benefits matter to them, and 4) whether they have sufficient support to make their treatment decision. We expanded items 2 and 3 into four separate items assessing risks and benefits individually. Responses were summed, resulting in a scale of 0-6, where 0 indicates maximum conflict and 6 indicates no conflict
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
Number analyzed (Participants) | 79 | 75
units on a scale | 5.2 (1.7) | 5.5 (1.2)

5. Secondary Outcome: Number of Participants Who Achieve Their Preferred Role in Treatment Decision Making Process
Description: Achievement of preferred role in decision-making was assessed by the Control Preferences Scale; patients indicate the role they played in their treatment decision which is compared to their preferred role (assessed at baseline).
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
Number analyzed (Participants) | 79 | 75
Participants
  No | 48 | 39
  Yes | 30 | 35
  Unknown/missing | 1 | 1

6. Secondary Outcome: Satisfaction When Making a Chemotherapy Treatment Choice: PACE Scores
Description: Satisfaction with communication during treatment decision-making process was assessed via 5 items from the Patient Assessment of Cancer Communication Experiences (PACE). Scores were averaged ("does not apply" excluded), creating a score of 1 to 4, with 4 being the most satisfied.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
Number analyzed (Participants) | 79 | 75
units on a scale | 3.6 (0.5) | 3.7 (0.4)

7. Secondary Outcome: Number of Participants Who Have End-of-life Discussions With Healthcare Proxy and Care Team
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
Number analyzed (Participants) | 71 | 73
Participants
  No | 60 | 55
  Yes | 10 | 16
  Unknown/missing | 1 | 2

8. Secondary Outcome: Decisional Regret When Making a Chemotherapy Treatment Choice: Decisional Regret Scale
Description: Decisional Regret was assessed at the 3-month survey using Brehaut's 5-item decisional regret scale, with scores ranging from 0-100, where 100 indicates maximal regret, and 0 indicates no regret.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
Number analyzed (Participants) | 71 | 73
units on a scale | 79.6 (19.3) | 84.7 (14.4)

9. Secondary Outcome: Emotional Distress When Making a Chemotherapy Treatment Choice: FACT-G Assessment
Description: Emotional distress was assessed via the emotional wellbeing subscale of the FACT-G. Scores range from 0-24, with higher scores being more desirable.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
Number analyzed (Participants) | 71 | 73
units on a scale | 16.5 (4.6) | 17.3 (4.5)

10. Secondary Outcome: Patient-Reported Prognostic Understanding in Median Years
Description: Prognostic understanding was assessed by asking patients about their understanding of the prognosis of the typical patient with their condition (<1 year, 1-2 years, 2- 3 years, 3-5 years, 5-10 years, >10 years). This measure was adapted from the CANCORS trial.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
Number analyzed (Participants) | 71 | 73
years | 2.5 [1.5 to 4.0] | 2.5 [1.5 to 4.0]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 months
Description: All participants were monitored for adverse events throughout their time on the study. On average, participants were involved in the trial for 3 months.
Arm/Group | Patient Usual Care Arm | Patient Investigational Care Arm
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/92
Other Adverse Events (participants affected / at risk) | 0/94 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT02282722/Prot_SAP_000.pdf